CLINICAL TRIAL: NCT00516074
Title: A Study to Assess the Effect of Exenatide Treatment on Mean 24-Hour Heart Rate in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-MC-GWCD
Record Dates: First submitted 2007-08-10; First posted 2007-08-14 (Estimated); Results first posted 2009-06-12 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exenatide; Byetta; type 2 diabetes; heart rate; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide Arm (Experimental): This arm will receive 5mcg exenatide for 4 weeks, and then 10mcg exenatide for the remaining 8 weeks of the study.
  Interventions: Drug: exenatide
- Placebo Arm (Placebo Comparator): This arm will receive placebo injection (volume equivalent to the exenatide injection in the experimental arm).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg or 10mcg, twice a day
  Other Names: Byetta; AC2993; LY2148568
  Arms: Exenatide Arm
Drug: placebo — subcutaneous injection, volume equivalent to active, twice a day
  Arms: Placebo Arm

SUMMARY:
This study will explore the effect of exenatide (given twice a day) versus placebo (given twice a day) treatment on change in mean 24-hour heart rate over a 12 week period of drug exposure in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes.
* Treated with metformin and/or a thiazolidinedione.
* HbA1c between 6.5% and 9.5%, inclusive.
* Body Mass Index (BMI) > 25 kg/m^2 and < 40 kg/m^2.

Exclusion Criteria:

* Have previously received exenatide or glucagon-like peptide-1 analogs.
* Have participated in an interventional medical, surgical, or pharmaceutical study (a study in which an experimental, drug, medical, or surgical treatment was given) within 30 days of screening. This criterion includes drugs that have not received regulatory approval for any indication at the time of study entry.
* Receiving beta blockers.
* Receiving treatment with a drug directly affecting gastrointestinal motility, including but not limited to Reglan® (metoclopramide), Propulsid® (cisapride), and chronic macrolide antibiotics.
* Have received treatment with systemic glucocorticoid therapy by oral, intravenous (IV), or intramuscular (IM) route within 6 weeks of screening, or are regularly treated with potent, inhaled intranasal steroids that are known to have a high rate of systemic absorption or bronchodilators.
* Have been treated with drugs that promote weight loss (for example, Adipex® [phentermine], Acomplia® [rimonabant], Xenical® [orlistat], Meridia® [sibutramine], Acutrim® [phenylpropanolamine], or similar over-the-counter medications) within 3 months of screening.
* Have been treated for longer than 2 weeks with any of the following excluded medications within 3 months prior to screening: *Insulin; *Alpha-glucosidase inhibitors (for example, Glyset® [miglitol] or Precose® [acarbose]); *Meglitinides (for example, Prandin® [repaglinide] or Starlix® [nateglinide]); *Sulfonylureas (for example, Glucotrol® [glipizide] or Micronase® [glyburide]); *Dipeptidyl peptidase IV (DPP-IV) inhibitors (for example, Januvia™ [sitagliptin])
* Have donated blood within 60 days of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (6):
- Canada (2):
  - Research Site, Halifax, Nova Scotia
  - Research Site, Toronto, Ontario
- Netherlands (4):
  - Research Site, Etten-Leur
  - Research Site, Leiden
  - Research Site, Rotterdam
  - Research Site, Utrecht

REFERENCES:
- [Derived] Gill A, Hoogwerf BJ, Burger J, Bruce S, Macconell L, Yan P, Braun D, Giaconia J, Malone J. Effect of exenatide on heart rate and blood pressure in subjects with type 2 diabetes mellitus: a double-blind, placebo-controlled, randomized pilot study. Cardiovasc Diabetol. 2010 Jan 28;9:6. doi: 10.1186/1475-2840-9-6. PMID 20109208

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide BID: 5mcg exenatide twice daily for 4 weeks, and then 10mcg exenatide twice daily for the remaining 8 weeks of the study.
- Placebo: Placebo injection twice daily (volume equivalent to the exenatide injection in the experimental arm).
Period: Overall Study
Arm/Group | Exenatide BID | Placebo
Started | 28 | 26
Completed | 22 | 23
Not Completed | 6 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Subject Decision | 4 | 2
Not completed — Loss of Glucose Control | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide BID | Placebo | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.62 (10.90) | 54.14 (10.13) | 55.43 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 19 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean 24-hour Heart Rate From Baseline to Endpoint
Description: Change from baseline to endpoint in average heart rate measured over 24 hours by an ambulatory blood pressure monitor.
Time Frame: 12 weeks
Population: Intent to treat; Last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 26 | 25
beats per minute
  Baseline (Week 0) | 74.83 (2.04) | 74.47 (2.08)
  Change at endpoint (Week 12) | 2.14 (1.39) | -0.71 (1.42)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Non-Inferiority or Equivalence — Approximately 25 subjects were intended to be randomized to both the exenatide and placebo arms. Assuming an approximate 24% dropout rate, 19 patients per treatment arm would complete the study. A sample of 19 patients per treatment group would provide 90% power to detect a 10 bpm difference between treatment groups in change in daily mean heart rate from baseline; p = 0.1585, ANCOVA

2. Secondary Outcome: Change in Daytime Heart Rate From Baseline to Endpoint
Description: Change from baseline to endpoint in daytime heart rate as measured by an ambulatory blood pressure monitor
Time Frame: 12 weeks
Population: Intent to treat; Last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 26 | 25
beats per minute
  Baseline (Week 0) | 75.97 (2.22) | 75.37 (2.26)
  Change at endpoint (Week 12) | 2.35 (1.59) | -0.87 (1.62)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Non-Inferiority or Equivalence — Power calculation for the primary endpoint is described as part of the primary endpoint information above; p = 0.1624, ANCOVA

3. Secondary Outcome: Change in Nighttime (2400-0600) Heart Rate From Baseline to Endpoint
Description: Change from baseline to endpoint in nighttime (2400-0600) heart rate as measured by an ambulatory blood pressure monitor
Time Frame: 12 weeks
Population: Intent to treat; Last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 26 | 25
beats per minute
  Baseline (Week 0) | 71.54 (2.12) | 71.77 (2.16)
  Change at endpoint (Week 12) | 1.43 (1.79) | -0.28 (1.83)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Non-Inferiority or Equivalence — Power calculation for the primary endpoint is described as part of the primary endpoint information above; p = 0.5077, ANCOVA

4. Secondary Outcome: Change in Mean 24 Hour Systolic Blood Pressure From Baseline to Endpoint
Description: Change from baseline to endpoint in average systolic blood pressure measured over 24 hours by an ambulatory blood pressure monitor
Time Frame: 12 weeks
Population: Intent to treat; Last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 26 | 25
mmHg
  Baseline (Week 0) | 126.61 (3.04) | 119.93 (3.10)
  Change at endpoint (Week 12) | -0.81 (2.67) | -0.34 (2.72)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Non-Inferiority or Equivalence — Power calculation for the primary endpoint is described as part of the primary endpoint information above; p = 0.9034, ANCOVA

5. Secondary Outcome: Change in Mean 24 Hour Diastolic Blood Pressure From Baseline to Endpoint
Description: Change from baseline to endpoint in average diastolic blood pressure measured over 24 hours by an ambulatory blood pressure monitor
Time Frame: 12 weeks
Population: Intent to treat; Last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 26 | 25
mmHg
  Baseline (Week 0) | 75.70 (2.05) | 70.54 (2.09)
  Change at endpoint (Week 12) | -0.60 (1.49) | -2.34 (1.52)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Non-Inferiority or Equivalence — Power calculation for the primary endpoint is described as part of the primary endpoint information above; p = 0.4270, ANCOVA

6. Secondary Outcome: Change in Hemoglobin A1c (HbA1c) From Baseline to Endpoint
Description: Change from baseline to endpoint in HbA1c
Time Frame: 12 weeks
Population: Intent to treat; Last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Exenatide BID | Placebo
Number analyzed (Participants) | 27 | 25
percent
  Baseline (Week 0) | 7.50 (0.16) | 7.11 (0.17)
  Change at endpoint (Week 12) | -0.15 (0.16) | 0.12 (0.17)
Statistical Analysis 1: Comparison: Exenatide BID vs Placebo; Test type: Non-Inferiority or Equivalence — Power calculation for the primary endpoint is described as part of the primary endpoint information above; p = 0.2600, ANCOVA

ADVERSE EVENTS:
Arm/Group | Exenatide BID | Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 1
Other Adverse Events (participants affected / at risk) | 18 | 21
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Exenatide BID | Placebo
Rib fracture (Injury, poisoning and procedural complications) | 1/28 | 0/26
Depression (Psychiatric disorders) | 0/28 | 1/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Exenatide BID | Placebo
Nausea (Gastrointestinal disorders) | 10/28 | 5/26
Headache (Nervous system disorders) | 5/28 | 4/26
Influenza (Infections and infestations) | 5/28 | 7/26
Cough (Respiratory, thoracic and mediastinal disorders) | 2/28 | 0/26
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2/28 | 1/26
Vomiting (Gastrointestinal disorders) | 2/28 | 2/26
Dizziness (Nervous system disorders) | 1/28 | 2/26
Hyperglycemia (Metabolism and nutrition disorders) | 1/28 | 5/26
Depression (Psychiatric disorders) | 0/28 | 2/26
Migraine (Nervous system disorders) | 0/28 | 2/26
Restlessness (Nervous system disorders) | 0/28 | 2/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days